CLINICAL TRIAL: NCT06227741
Title: Concept Mapping: as a Tool for Problem Based Learning on Students Problem Solving Skills, Metacognitive Awareness, and Self-directed Learning
Brief Title: Concept Mapping: as a Tool for Problem Based Learning
Acronym: ConceptMapp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB0001260
Record Dates: First submitted 2023-12-25; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-12

CONDITIONS: Educational Problems; Problem;Learning
Keywords: education; concept mapping; Problem Solving skills

STUDY DESIGN:
Intervention Model Description: concept mapping
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concept mapping (Experimental): utility of concept mapping as a learning tool for problem solving. As well, examine the effect of using concept mapping as a tool for problem based learning on students' Metacognitive Awareness, problem solving skills, , and self -directed learning at Zagazig Faculty of Nursing
  Interventions: Other: Concept Mapping: as a Tool for Problem Based Learning
- traditional learning experience (No Intervention): utility of traditional learning experience as a learning tool

INTERVENTIONS:
Other: Concept Mapping: as a Tool for Problem Based Learning — Concept mapping is a visual representation and organizational tool that illustrates the relationships between concepts, ideas, and information. It involves creating a graphical depiction of knowledge, typically using nodes or boxes to represent concepts and connecting lines or arrows to signify the relationships between them. The central concept or main idea is often positioned in the center of the map, with subsidiary concepts branching out from it. These maps serve as a comprehensive overview of a subject, highlighting the hierarchical structure and interconnectedness of various elements.
  Arms: concept mapping

SUMMARY:
This study delves into the utilization of concept mapping as a strategic tool within problem-based learning (PBL) to enhance students' problem-solving skills, metacognitive awareness, and self-directed learning abilities. Concept mapping, a visual representation of knowledge structures, is explored as a means to cultivate and refine students' problem-solving capabilities, preparing them for challenges in various domains.

DETAILED DESCRIPTION:
This study delves into the utilization of concept mapping as a strategic tool within problem-based learning (PBL) to enhance students' problem-solving skills, metacognitive awareness, and self-directed learning abilities. Concept mapping, a visual representation of knowledge structures, is explored as a means to cultivate and refine students' problem-solving capabilities, preparing them for challenges in various domains. Additionally, the research investigates how concept mapping within a PBL context promotes metacognitive awareness, helping students become more conscious of their learning strategies and enabling them to identify gaps in understanding. Moreover, the study explores the role of concept mapping in empowering self-directed learning, fostering autonomy and a deeper sense of ownership over students' educational journeys. The insights gained from this research not only inform instructional design practices, providing evidence-based strategies for enhancing problem-based learning through concept mapping but also contribute to the broader educational research discourse, offering valuable perspectives on effective teaching and learning strategies.

ELIGIBILITY:
Inclusion Criteria:

* from 2 -4th academic year
* accept to participate in this study

Exclusion Criteria:

* first academic year
* psychological or mental disorder

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
improving students' metacognitive awareness | 2 months
  Nursing students exposed to the concept mapping technique exhibited a higher score in the metacognitive awareness skills inventory ( total scores ranging from 30: 150 and a higher score of more than 90 indicating higher Metacognitive Awareness) than those not exposed to concept mapping.
improving students' Problem-Based Learning | 2 months
  Nursing students exposed to the concept mapping technique exhibited a higher score on the problem-solving skills questionnaire( total scores range from 28 to 140 and higher scores more than 56 indicating higher problem-solving skills) than students not exposed to concept mapping.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H atta, Study Chair — Faculty of nursing, Alexandria university, Egypt
Locations (1):
- Faculty of Nursing, Masjid al Khiḑr, Semoha, Egypt

DOCUMENTS (1):
  • Study Protocol (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT06227741/Prot_000.pdf